CLINICAL TRIAL: NCT01535365
Title: Heat Versus Ice in the Acute Management of Neck and Back Strain Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Adam Singer, md, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20076955
Record Dates: First submitted 2010-11-05; First posted 2012-02-17 (Estimated); Results first posted 2012-02-17 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Back Strain; Neck Strain
Keywords: muscular sprain; acute back pain; acute neck pain; heat treatment; cold treatment
MeSH Terms: conditions — Fever | interventions — Hot Temperature; Cold Temperature

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Heat (Active Comparator): Application of Heat pad to site of muscle sprain.
  Interventions: Other: Heat
- Cold (Active Comparator): Application of ice pack to muscle sprain.
  Interventions: Other: Cold

INTERVENTIONS:
Other: Heat — Application of heat pack to the back or neck sprain.
  Other Names: warm pack
  Arms: Heat
Other: Cold — Application of ice pack to the back or neck sprain.
  Arms: Cold

SUMMARY:
Muscle sprains of the back and neck are very common. In addition to pain and antiinflammatory medications the use of either cold or hot packs has been recommended. In the current study we will compare ice packs and heat packs to see which is more effective at relieving pain from back and neck sprains while in the Emergency Department.

DETAILED DESCRIPTION:
as above

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients with acute neck or back pain who are able to consent and are in pain on arrival to Emergency Department.

Exclusion Criteria:

* Those unable or unwilling to consent, those with suspected fractures or neurologic deficits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-03; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ADAM SINGER, MD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University Medical Center, Stony Brook, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Heat: Application of Heat to site of muscle sprain.
- Cold: Application of cold to muscle sprain.
Period: Overall Study
Arm/Group | Heat | Cold
Started | 31 | 29
Completed | 31 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Heat | Cold | Total
Number analyzed (Participants) | 31 | 29 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0.0
  Between 18 and 65 years | 31 | 29 | 60.0
  >=65 years | 0 | 0 | 0.0
Age Continuous [Mean (Standard Deviation); unit: years] | 37.8 (14.7) | 36.3 (11.2) | 37.1 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31.0
  Male | 15 | 14 | 29.0
Region of Enrollment [Number; unit: participants]
  United States | 31 | 29 | 60.0

OUTCOME MEASURES:

1. Primary Outcome: Pain Score After Treatment
Description: Pain measured with validated 100 mm VAS with 0 representing no pain and 100 representing most severe pain imaginable
Time Frame: 30 minutes
Population: this sample size gives 80% power to detect a size effect of one SD
Measure: Mean (95% Confidence Interval); unit: mm
Groups:
- Heat Pack: Application of Heat to site of muscle sprain.
- Ice Pack: Application of cold to muscle sprain.
Arm/Group | Heat Pack | Ice Pack
Number analyzed (Participants) | 31 | 29
mm | 66 (16) [57 to 75] | 64 (10) [56 to 73]

2. Secondary Outcome: Request for Rescue Analgesia
Description: Number of participants requesting a rescue analgesic be given
Time Frame: 30 minutes
Measure: Number; unit: Participants
Arm/Group | Heat | Cold
Number analyzed (Participants) | 31 | 29
Participants | 18 | 12

ADVERSE EVENTS:
Arm/Group | Heat | Cold
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/29
Other Adverse Events (participants affected / at risk) | 0/31 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes